CLINICAL TRIAL: NCT07018843
Title: Metabolic Characterisation of Critically Ill Patients: An Observational Study Focusing on Mitochondria
Brief Title: Mitochondrial Assessment in Critical Ill Patients in Intensive Care
Acronym: MitoICU
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM CRI0453
Record Dates: First submitted 2025-01-23; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-01

CONDITIONS: Critical Illness
Keywords: Mitochondria; Critical illness; Respirometry; Muscle biopsy; Breath test; Oroboros; MyotonPRO; Muscle ultrasound
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Platelet specimens
  2. Muscle biopsy specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Critically unwell intubated adults on ICU: The participants must be over 18, recruited within 48-hours of intubation and likely to remain intubated and ventilated for > 72-hours.

SUMMARY:
Critically ill patients often require admission to the intensive care unit (ICU). When patients develop organ failures and end up on a ventilator, there are changes in the body's cell function that can increase the risk of poor outcomes. All cells, in order to function normally, have mitochondria, which help them generate energy and transfer vital messages between cells. However, during critical illness, the mitochondria in the cells can function less effectively and die prematurely, or their new synthesis and regeneration can be severely affected. This can result in continuous multi-organ failure with a lack of recovery and muscle wasting, causing severe weakness and an inability to function normally.

In this study, the investigators aim to assess mitochondrial capacity using three methods with varying levels of invasiveness. The investigators are planning to recruit 20 patients in the ICU who are on a ventilator for breathing support. The investigators plan to measure mitochondrial capacity from a breath test, blood cells, and muscle cells.

The investigators will collect breath samples after consuming an amino acid, which is a component of protein in our body and is commonly found in food. This amino acid is only broken down by the mitochondria. This safe test allows us to measure how much mitochondrial capacity remains in the body after the modified amino acid is broken down by the mitochondria. In comparison, the investigators will use standard methods which includes blood tests and muscle biopsy to examine the mitochondrial function of platelets (blood cells) and muscle cells. The investigators will also use non-invasive techniques (ultrasound and 'MyotonPRO') to assess muscle.

This study will help us determine the best way to assess mitochondrial function and capacity in critically ill patients and to understand strengths and weaknesses of different approaches.

When patients' mitochondrial function or capacity is impaired, the investigators can provide them with particular nutrition to improve mitochondrial activity. Because evaluating this at the bedside is challenging, it is impossible to tell which patients may benefit from specific therapies that improve mitochondrial function. If this breath test provides an assessment similar to the standard, sophisticated mitochondrial testing, the investigators could use it at the bedside in the future, which may improve patient outcomes and help design large clinical trials.

DETAILED DESCRIPTION:
Critical illness is associated with significantly increased risk of morbidity and mortality (Morgan, 2021). Patients are often admitted to the intensive care unit (ICU) with single or multiple organ failure of diverse aetiology (e.g., severe infection, inflammation, trauma). Multi-organ failure is related to cellular and bioenergetic dysfunction caused by hypoxia, hyperoxia and increased oxidative stress and despite organ support measures, the anticipated mortality is high with ~20-50% (Zambon and Vincent, 2008). Despite these negative consequences, therapeutic strategies are limited with nearly all ICU based clinical studies failing to identify treatments that improve clinical outcomes. The heterogeneity within the ICU patients coupled with the lack of phenotypic characterisation has contributed to this poor progress, highlighting the need to comprehensively characterise the ICU phenotype to develop effective interventions that improve clinical outcomes.

Mitochondria have vital functions beyond cellular energy metabolism, including regulating cell death, calcium homeostasis and modulation of the cell cycle. All of these functions have been shown to impact outcomes during critical illness with mitochondria exhibiting structural changes within days of being admitted to ICU (Klawitter et al., 2023). Despite appropriate ICU management with antibiotics, fluids, oxygenation and nutrition, sepsis- associated mortality remains high and this is thought to be due to persistence of inflammation and impaired mitochondrial processes (Supinski et al, 2020). Stressed mitochondria produce higher levels of reactive oxygen species, activating caspases, and triggering cell death. Following mitochondrial death, subsequent lack in ATP production has been suggested to lead to poor clinical outcomes. Mitochondrial death itself leads to poor clinical outcomes and a study in 2013 directly linked higher levels of circulating mtDNA to increased ICU mortality at 28-days post admission (Jameson et al., 2023).

Physical inactivity is strongly associated with alterations in mitochondrial dysfunction and consequently prolonged inactivity in ICU may lead to adverse outcomes. Studies show downregulation of key mitochondrial transcription factors in skeletal muscle even in early stages of critical illness (Klawitter et al., 2023). A recent randomised control trial concluded that there was persistent intramuscular inflammation in critical illness and demonstrated that exercise alone is insufficient to restore muscle function (Jameson et al., 2023). A defining feature of ICU patients is the rapid and substantial loss of muscle (Puthucheary et al., 2023), which significantly increases morbidity and mortality risk (key clinical outcomes of ICU) (Lee et al., 2021).

Associated with ICU induced muscle decline is mitochondrial dysfunction, characterised by reduced mitochondrial content and function (Puthucheary et al., 2018). However, where mitochondrial deficiencies occur (e.g., which complex of the electron transport chain), and thus which element of the mitochondria are best to target therapeutically to improve mitochondrial health remains' elusive. These fundamental questions can be addressed using sophisticated omic-informatic techniques; however, this system biology approach requires interdisciplinary expertise, which has stunted progress. Bridging this gap, the investigators have interdisciplinary expertise in applying advanced computational analysis to human biological samples, permitting the detection of molecular targets to improve muscle mitochondrial health (Deane et al., 2019; Deane et al., 2023; Deane et al., 2021). Thus, using our pipeline, it is possible to identify molecular regulators of, and promising interventional avenues for, improving mitochondrial health in ICU patients.

Monitoring mitochondrial function in patients is a bedside challenge, as it requires muscle biopsies followed by laboursome laboratory processing and analysis. Therefore, there is an unmet need to develop minimally or non-invasive methods to assess mitochondrial function to aid clinical decision-making processes. Addressing this research gap, the investigators have developed a novel isotope labelled non-invasive breath test to evaluate mitochondrial function rapidly and repeatedly, which has been validated in healthy subjects and in patients with non-alcoholic fatty liver disease (Afolabi et al., 2018).

Emerging pilot data from healthy and clinical (elective surgery) cohorts demonstrating our inhouse ability to perform mitochondrial functional assessment in muscle tissue and platelets using the Oroboros, and via the breath test using mass spectrometry. However, the correspondence between the measures and the applicability in ICU patients remains to be determined. Taken together and based on our pilot data, the investigators strongly believe it is feasible to take complementary mitochondria-focussed metabolic and molecular measurements in ICU patients, to better characterise ICU cohorts and identify future therapeutic avenues. By using a multitude of different strategies to assess mitochondrial capacity the investigators aim to better understand how it is affected in critical illness on both a systemic and tissue level.

One emerging and promising approach is the use of 13C-breath tests (13C-BTs) to characterise mitochondrial capacity. 13C-BTs involves the oral administration of a metabolic substrate labelled with a non-radioactive stable isotope of carbon (13C-atom), which is metabolised exclusively within the mitochondria and is followed by the recovery of the 13C-tracer on the breath as 13CO2. The 13C-substrate can be chosen to evaluate mitochondrial metabolism in the whole body. An example of a 13C-BT is the 13C-ketoisocaproate breath test (13C-KICA BT) which assesses mitochondrial function. It involves the oral ingestion of 13C-KICA, a metabolic intermediate of the branched chain amino acid leucine, which is metabolised in the mitochondria to 13C-labelled carbon dioxide (13CO2) which is recovered on the breath of the subject (Afolabi et al., 2018). This pathway is catalysed by the branched chain alpha-ketoacid dehydrogenase, which is in the mitochondria over a period of time. Thus, the generation of 13CO2 following the oral administration of 13C-KICA should reflect mitochondrial metabolism.

The ability to monitor changes in mitochondrial metabolism in patients with critical illness at an early stage is crucial, to develop effective approaches to treat patients early. This novel non-invasive method of assessing mitochondrial capacity has the potential to use at the bedside to inform treatment decisions.

There is an urgent need for practical, sensitive tests of metabolic function that can help to identify potential therapeutic targets in critical illness and quantify mitochondrial dysfunction.

Non-invasive 13C-breath tests such as the 13C-ketoisocaproate (13C-KICA) breath test can give a rapid quantitative measure of whole-body mitochondrial capacity providing invaluable information regarding the patients' metabolic function at any given point in time. Thus, allowing the evaluation of the response to targeted therapies.

Hypothesis of MitoICU: Mitochondrial capacity can be assessed in critically ill patients from multiple compartments (whole body and liver: 13C-KICA; cellular: platelets; and tissue: skeletal muscle) and the non-invasive measures (muscle ultrasound and MyotonPRO) may be used as surrogate for mitochondrial assessment in ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* Mechanically ventilated at time of recruitment
* Defined as critically ill by the responsible clinician
* Recruited within 48-hours of intubation
* Likely to remain intubated and ventilated for > 72-hours

Exclusion Criteria:

* Patients < 18 years
* Patient is being treated on an end-of-life pathway or active treatment is likely to be withdrawn within 24-hours
* Patient has significant liver dysfunction (Child-Pugh ≥ class 3)
* Patient is not absorbing enterally (defined as 2 x NG aspirates of > 500ml)
* Known pregnancy or positive urinary pregnancy test on testing
* Specific exclusion criteria for the muscle biopsy component of the study: Patients taking treatment dose anticoagulation, antiplatelet agents or with severe coagulopathy (or disease process leading to increased risk of bleeding) will be excluded from having a muscle biopsy taken as part of data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult (>18 years) patients who have been mechanically ventilated will be recruited from the Intensive Care Unit at University Hospital Southampton.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of assessing mitochondrial capacity by three different methods | 15 months
  Feasibility of assessing mitochondrial capacity in critically ill patients from different biological samples [skeletal muscle, platelets and breath] by three different methods, assessing the proportion of successful participants recruited, samples taken, and samples processed. The physiologic parameter used to assess each of these methods is detailed further below.

SECONDARY OUTCOMES:
To evaluate mitochondrial capacity using 13C-ketoisocaproate breath test. | 15 months
  To evaluate the mitochondrial capacity in critically ill patients using the 13C-ketoisocaproate breath test. Data collection is in the form of breath samples taken from the ventilator circuit. Exhaled ratio of 13CO2 following the oral administration of 13C-KICA should reflect mitochondrial metabolism and is used to assess the outcome measure.
To evaluate mitochondrial capacity using mitochondrial respiration in skeletal muscle | 15 months
  To evaluate global mitochondrial capacity in critically ill patients using mitochondrial respiration in skeletal muscle. Muscle samples will be assessed using high resolution respirometry to assess their mitochondrial capacity and function.
To evaluate mitochondrial capacity using the mitochondrial respiration of platelets | 15 months
  To evaluate mitochondrial capacity by measuring the mitochondrial respiration of platelets in critically ill patients. Mitochondrial capacity and function of platelets will be assessed using high resolution respirometry, to allow assessment of this outcome measure.
Longitudinal assessment of mitochondrial capacity in critical illness | 15 months
  Longitudinal assessment of mitochondrial capacity in critical ill patients during their admission to critical care. The physiological parameters described in the other objectives of this study will be assessed over 120 hours to assess how mitochondrial function may change over this period.
Comparison of mitochondrial capacity across the secondary outcome measures. | 15 months
  Comparing platelet (systemic) mitochondrial capacity with skeletal muscle (tissue) mitochondrial capacity and global body mitochondrial capacity (C-KICA). The physiological parameters described in the other objectives of this study will be compared to assess the ways these outcomes reflect mitochondrial capacity and function.

OTHER OUTCOMES:
Exploratory outcome 1: To assess targeted and untargeted metabolomics in critically ill patients using analysis of the metabolites in biological samples collected. | 15 months
  To assess targeted and untargeted metabolomics in critically ill patients. This outcome measure will be assessed using analysis of the samples collected (blood and muscle).
Exploratory outcome 2: To assess mitochondrial specific metabolic markers in critically ill patients | 15 months
  The outcome will be assessed using redox analysis of the samples collected.
Exploratory outcome 3: To assess oxidative stress in critically ill patients | 15 months
  The outcome will be assessed using redox analysis of the samples collected.
Exploratory outcome 4: To assess redox variations in critically ill patients | 15 months
  The outcome will be assessed using redox analysis of the samples collected.
Exploratory outcome 5: To assess fatty acid profiles of red cells in critically ill patients | 15 months
  The outcome will be assessed using redox analysis of the samples collected.
Exploratory outcome 6: To assess the clinical outcomes of the patients within the study | 15 months
  This outcome measure will be assessed by collecting clinical information regarding the patient outcomes in the study including duration of mechanical ventilation, duration of ICU and hospital length of stay, ICU and hospital mortality.
Exploratory outcome 7: To assess muscle health status and echogenicity (using ultrasound imaging) during critical illness | 15 months
  Muscle thickness measurements and cross-sectional area will be taken from the right side of rectus femoris and vastus intermedius, vastus lateralis and biceps brachii. Muscle echogenicity will be measured using ultrasound imaging of quadriceps, including rectus femoris and vastus lateralis.
Exploratory outcome 8: To assess muscle using the MyotonPRO device during critical illness | 15 months
  The myotonPRO device assesses muscle elasticity, stiffness and tone. Measurements will be taken from rectus femoris, vastus lateralis, and biceps brachii, at locations described in the ultrasound section above. With tone (Hz), dynamic stiffness (N/m) and elasticity (logarithmic decrement; log) measurements taken.

CONTACTS AND LOCATIONS:
Overall Officials: Ahilanandan Dushianthan, MBBS MRCP PhD, Principal Investigator — University of Southampton; University Hospital Southampton
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afolabi PR, Scorletti E, Smith DE, Almehmadi AA, Calder PC, Byrne CD. The characterisation of hepatic mitochondrial function in patients with non-alcoholic fatty liver disease (NAFLD) using the 13C-ketoisocaproate breath test. J Breath Res. 2018 Jul 19;12(4):046002. doi: 10.1088/1752-7163/aacf12. PMID 29943733
- [Background] Deane CS, Willis CRG, Phillips BE, Atherton PJ, Harries LW, Ames RM, Szewczyk NJ, Etheridge T. Transcriptomic meta-analysis of disuse muscle atrophy vs. resistance exercise-induced hypertrophy in young and older humans. J Cachexia Sarcopenia Muscle. 2021 Jun;12(3):629-645. doi: 10.1002/jcsm.12706. Epub 2021 May 5. PMID 33951310
- [Background] Deane CS, Phillips BE, Willis CRG, Wilkinson DJ, Smith K, Higashitani N, Williams JP, Szewczyk NJ, Atherton PJ, Higashitani A, Etheridge T. Proteomic features of skeletal muscle adaptation to resistance exercise training as a function of age. Geroscience. 2023 Jun;45(3):1271-1287. doi: 10.1007/s11357-022-00658-5. Epub 2022 Sep 26. PMID 36161583
- [Background] Deane CS, Ames RM, Phillips BE, Weedon MN, Willis CRG, Boereboom C, Abdulla H, Bukhari SSI, Lund JN, Williams JP, Wilkinson DJ, Smith K, Gallagher IJ, Kadi F, Szewczyk NJ, Atherton PJ, Etheridge T. The acute transcriptional response to resistance exercise: impact of age and contraction mode. Aging (Albany NY). 2019 Apr 15;11(7):2111-2126. doi: 10.18632/aging.101904. PMID 30996129
- [Background] Puthucheary ZA, Astin R, Mcphail MJW, Saeed S, Pasha Y, Bear DE, Constantin D, Velloso C, Manning S, Calvert L, Singer M, Batterham RL, Gomez-Romero M, Holmes E, Steiner MC, Atherton PJ, Greenhaff P, Edwards LM, Smith K, Harridge SD, Hart N, Montgomery HE. Metabolic phenotype of skeletal muscle in early critical illness. Thorax. 2018 Oct;73(10):926-935. doi: 10.1136/thoraxjnl-2017-211073. Epub 2018 Jul 6. PMID 29980655
- [Background] Lee ZY, Ong SP, Ng CC, Yap CSL, Engkasan JP, Barakatun-Nisak MY, Heyland DK, Hasan MS. Association between ultrasound quadriceps muscle status with premorbid functional status and 60-day mortality in mechanically ventilated critically ill patient: A single-center prospective observational study. Clin Nutr. 2021 Mar;40(3):1338-1347. doi: 10.1016/j.clnu.2020.08.022. Epub 2020 Aug 28. PMID 32919818
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Jameson TSO, Caldow MK, Stephens F, Denehy L, Lynch GS, Koopman R, Krajcova A, Urban T, Berney S, Duska F, Puthucheary Z. Inflammation and altered metabolism impede efficacy of functional electrical stimulation in critically ill patients. Crit Care. 2023 Nov 6;27(1):428. doi: 10.1186/s13054-023-04664-7. PMID 37932834
- [Background] Supinski GS, Schroder EA, Callahan LA. Mitochondria and Critical Illness. Chest. 2020 Feb;157(2):310-322. doi: 10.1016/j.chest.2019.08.2182. Epub 2019 Sep 5. PMID 31494084
- [Background] Klawitter F, Ehler J, Bajorat R, Patejdl R. Mitochondrial Dysfunction in Intensive Care Unit-Acquired Weakness and Critical Illness Myopathy: A Narrative Review. Int J Mol Sci. 2023 Mar 14;24(6):5516. doi: 10.3390/ijms24065516. PMID 36982590
- [Background] Zambon M, Vincent JL. Mortality rates for patients with acute lung injury/ARDS have decreased over time. Chest. 2008 May;133(5):1120-7. doi: 10.1378/chest.07-2134. Epub 2008 Feb 8. PMID 18263687
- [Background] Morgan A. Long-term outcomes from critical care. Surgery (Oxf). 2021 Jan;39(1):53-57. doi: 10.1016/j.mpsur.2020.11.005. Epub 2020 Dec 17. PMID 33519011